CLINICAL TRIAL: NCT04643223
Title: Effect of Elastic Bandage With Tension on the Inflammatory Response of Hypertrophic Scars in Patients With Deep Burns: a Randomized Triple Blind Trial
Brief Title: Effect of Elastic Bandage With Tension on the Inflammatory Response of Hypertrophic Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Fernando Figueira Integral Medicine Institute (Other)
Responsible Party: Principal Investigator, Alex Sandro Rolland de Souza, Prof. of IMIP's Stricto Sensu Post-graduation; Prof. Adjunct of the Federal University of Pernambuco; Prof. of the Catholic University of Pernambuco (UNICAP), Professor Fernando Figueira Integral Medicine Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: U1111-1231-9216
Record Dates: First submitted 2019-04-16; First posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Burns; Hypertrophic Scar
Keywords: burns; therapeutic elastic bandaging; functional bandage; Kinesio adhesive tapes; hypertrophic scar
MeSH Terms: conditions — Burns; Cicatrix, Hypertrophic | interventions — Athletic Tape

STUDY DESIGN:
Intervention Model Description: Clinical trial randomized triple blind sham controlled. An experimental group that will use the elastic bandage with seventy to ninety percent tension on the hypertrophic scar. It was a controlled sham that had used the elastic bandage without strain on the hypertrophic scar.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: This process will only be known to the researcher responsible for the project that will apply the kinesio tape on the scars; guaranteeing the concealment of the allocation with the triple masking, since the patients, the evaluators responsible for the Vancouver evaluation, the analysis of the histological and immunohistochemical material and the statistic will not be aware of this process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio tape with tension (Active Comparator): The intervention group will receive the elastic bandage - kinesio tape with tension between seventy to ninety percent on the selected hypertrophic scar. The application of kinesio tape follows a protocol, which involves the cleaning of the selected scar with liquid soap, drying, alcohol application for sebum removal, scar measurement and marking of the therapeutic zone and anchors. Following the application of the kinesio tape, with tension between seventy to ninety percent on the treated hypertrophic scar. This process follows the routine of patient care established by the service and will continue for a period corresponding to three months. In which, the Vancouver assessments and collections of scarring material for the histopathology will be carried out, in the time intervals corresponding to the beginning of the study intervention / entry (time 0), 45 days and 90 days after being eligible, to agree to participate in the study study and intervention.
  Interventions: Other: kinesio tape with tension
- Kinesio tape without tension (Sham Comparator): The controlled sham group will receive the application of kinesio tape without tension will follow the same protocol above, including the three moments of evaluation, beginning of the intervention (time 0), 45 days and 90 days, after the beginning of the intervention.
  Interventions: Other: kinesio tape without tension

INTERVENTIONS:
Other: kinesio tape with tension — The application of kinesio tape follows a protocol, which involves the sanitization of the selected scar with liquid soap, drying and application of alcohol to remove sebum. Measurement of the scar and marking of the therapeutic zone and anchors. Following the application of kinesio tape, with tension between seventy to ninety percent on the treated hypertrophic scar. This process follows the routine of patient care established by the service and will continue for a period corresponding to three months. In which, the evaluations of Vancouver, the collections of cicatricial material will be carried out, in the time spaces corresponding to forty-five and ninety days, having as reference the initial evaluation made after being elected.
  Other Names: Kinesio sport
  Arms: Kinesio tape with tension
Other: kinesio tape without tension — The application of kinesio tape without tension follows a protocol, which involves the sanitization of the selected scar with liquid soap, drying and application of alcohol to remove sebum. Measurement of the scar and marking of the therapeutic zone and anchors. Following application of the kinesio tape, no tension on the treated hypertrophic scar. This process follows the routine of patient care established by the service and will continue for a period corresponding to three months. In which, the evaluations of Vancouver, the collections of cicatricial material will be carried out, in the time spaces corresponding to forty-five and ninety days, having as reference the initial evaluation made after being elected.
  Other Names: Kinesio sport
  Arms: Kinesio tape without tension

SUMMARY:
Burns can lead to lesions of total thickness, which extend the reticular layer of the dermis requiring a healing process, resulting in aesthetic problems, hypertrophic and functional scars that causes the patient a state of low esteem and social isolation. Elastic bandage - Kinesio tape - is a low cost therapeutic resource when compared to the compression mesh and silicone gel plates, commonly indicated for the conservative treatment of these scars. The compressive effect of the bandage on the hypertrophic scar tissue promotes the reduction of local vascularization and the realignment of the collagen fibers, resulting in the repair of the multidirectional mobility of the treated tissue. The aim of the study is to determine the effect of elastic bandage with tension on the inflammatory response of hypertrophic scars in patients with deep burns. It is a randomized, triple blind study. Patients aged 18-59 years with hypertrophic scars due to burns will be included, and those with scaling and open wounds in scar tissue will be included, pregnant women and patients who have previously used any therapeutic resource that may have altered the remodeling process of the hypertrophic scar. The bandage will be applied on the scar selected by lottery. The intervention group will receive the bandage with a tension around 70% and the group will control the same bandage without tension. This feature will be used for a period of three to four days. Initial and subsequent evaluations will be performed after 45 and 90 days. Primary outcome: analysis of the inflammatory response. Through immunohistochemistry and the histological evaluation of the organization pattern of collagen fibers. Secondary: aesthetic and functional evaluation of the hypertrophic scar through the Vancouver scale. The statistical analysis will be done by the researcher and his collaborators, in addition to the statistical one, using the statistical programs Epi-Info 3.5 and Medcalc. For categorical variables, where appropriate, use of the chi-square test of association and Fisher's exact test. Regarding the quantitative variables, the unpaired samples were Student's t-test and if the distribution is not normal, the Mann-Whitney test will be used.

DETAILED DESCRIPTION:
Burns can lead to lesions of total thickness, which extend the reticular layer of the dermis requiring a repair process 1-2. This healing process, generally due to external and internal stimuli, causes scarring changes, among them, the hypertrophic scar 3-4. They develop about two months after the burn, occur more frequently in areas of high tension, preferably in the extensor faces of the joints or when they cross perpendicularly the lines of force of the skin. They exhibit scar tissue growth above the surface of the skin, respecting the limits of the original wound and are characterized by their reddish color, high stature, decreased flexibility and altered sensitivity 5-10. Patients with this type of scar can present stiffness in scar tissue, disfigurement, joint contractures, reduced range of motion, difficulties in daily functions and even psychological problems 11.

Mechanical strengths, when applied externally, can decrease the thickness of the epidermis, reduce the inflammatory response and promote a reorganization of the collagen fibers contained in the dermis, and thus improve the appearance of the vascularization and flexibility of the hypertrophic scar. Based on this principle, one of the therapeutic resources that can exert this external compressive effect is the elastic bandage - kinesio tape 12-13.

The use of elastic bandage - kinesio-taping is based on the principles of kinesiology and the self-healing ability of the organism. It takes advantage of the physical and mechanical properties of the bandage and the therapeutic action by the specific method of its application. Improving the appearance and perception of the scar, reducing functional limitations, thus repairing the patient's self-esteem 14-15.

Due to the few publications on the mechanism of action of elastic bandage, and its benefits, in the treatment of cicatricial sequelae due to burn. There was interest in seeking evidence that could support the mechanism of action of this therapeutic resource, and thus, a randomized, triple blind, controlled sham clinical trial was developed. It will be held at the Rehabilitation Center of the Governador Paulo Guerra Restoration Hospital (HR) located in Brazil and reference in the care of the burned patient. The study period will be from March 2018 to March 2020, with collection expected for June 2019 to November 2019.

The study population is the patients with hypertrophic scarring in the rehabilitation clinic of the HR. Patients will be picked up at the reception of this service, and they will be referred to the researcher responsible for the project. Once identified, the checklist of eligibility criteria and if eligible, patients will be invited by the researcher to participate in the study. In case of acceptance, the Informed Consent Form will be read aloud and if they agree to participate, they will sign it.

Those selected will be referred for initial clinical evaluation and other protocols that involve the study, among them, the selection of the scar, which will obey the inclusion criteria, and define the lesion treated with kinesio tape. In sequence, participants will be allocated randomly and stealthily through a computerized algorithm according to a table of sequential numbers from 1 to 30 using software R version 2.5.1. Generating the list of random allocation order, patients will use the letters A and B not knowing their meaning, being established only as treated with tension or without tension. Randomization is simple in two groups, the experimental or intervention group that will receive the kinesio tape with tension between seventy to ninety percent and the sham group with zero tension.

Patients will be referred for evaluation of the functional and aesthetic aspect of the hypertrophic scar, using as instrument of the Vancouver scale. In sequence will be taken to collect the scar material studied, through a biopsy performed at the Center for Treatment of Burns HR. After data collection, evaluation and biopsy, the treatment of patients is started. The therapeutic proposal will follow the routine of the service and the therapeutic protocol of the study common to all patients with cicatricial sequelae consisting of lubrication and massage of the scar and performing active free exercises and stretching for the limbs involved in the injury. It follows with the application of kinesio tape in the patients involved in the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Hypertrophic scars resulting from deep burns located in the upper and lower limbs and the anterior and posterior trunk;

Exclusion Criteria:

* Scar tissue showing scaling, somatosensory changes (touch, pressure and pain) and open wounds
* Pregnant women

Ages: 19 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
Histological pattern of the organization of the collagen fibers collected from the scar tissue (basal) | 0 day
  the evaluations will only be carried out in a descriptive qualitative way, since the histology is characterized by analysis of the cells together with their cell matrix. Thus the organization of the collagen fibers will be described as being distributed in parallel to the reticular layer of the dermis, or may also be described as randomly distributed to the reticular layer of the dermis. Characterizing a variable of type yes/no.
Histological pattern of the organization of the collagen fibers collected from the scar tissue (45o. day) | 45 days
  the evaluations will only be carried out in a descriptive qualitative way, since the histology is characterized by analysis of the cells together with their cell matrix. Thus the organization of the collagen fibers will be described as being distributed in parallel to the reticular layer of the dermis, or may also be described as randomly distributed to the reticular layer of the dermis. Characterizing a variable of type yes/no.
Histological pattern of the organization of the collagen fibers collected from the scar tissue (90o. day) | 90 days
  the evaluations will only be carried out in a descriptive qualitative way, since the histology is characterized by analysis of the cells together with their cell matrix. Thus the organization of the collagen fibers will be described as being distributed in parallel to the reticular layer of the dermis, or may also be described as randomly distributed to the reticular layer of the dermis. Characterizing a variable of type yes/no.

SECONDARY OUTCOMES:
Inflammatory response through immunohistochemistry (basal) | 0 day
  they correspond to the number of neutrophils, lymphocytes and mast cells that will be identified in the cicatricial tissue collected and analyzed quantitatively through the solft GRIMP 2.6. Where the amount of pixels emitted will be based on the color reaction pixel: brown (neutrophil), yellow (lymphocyte) and blue (mast cell). The program converts the pixel quantity of each color to a numerical value (n = Xμm). The analysis will be performed by a professional from the Ageu Magalhães Institute of the Federal University of Pernambuco.
Inflammatory response through immunohistochemistry (45o. day) | 45 days
  they correspond to the number of neutrophils, lymphocytes and mast cells that will be identified in the cicatricial tissue collected and analyzed quantitatively through the solft GRIMP 2.6. Where the amount of pixels emitted will be based on the color reaction pixel: brown (neutrophil), yellow (lymphocyte) and blue (mast cell). The program converts the pixel quantity of each color to a numerical value (n = Xμm). The analysis will be performed by a professional from the Ageu Magalhães Institute of the Federal University of Pernambuco.
Inflammatory response through immunohistochemistry (90o. day) | 90 days
  they correspond to the number of neutrophils, lymphocytes and mast cells that will be identified in the cicatricial tissue collected and analyzed quantitatively through the solft GRIMP 2.6. Where the amount of pixels emitted will be based on the color reaction pixel: brown (neutrophil), yellow (lymphocyte) and blue (mast cell). The program converts the pixel quantity of each color to a numerical value (n = Xμm). The analysis will be performed by a professional from the Ageu Magalhães Institute of the Federal University of Pernambuco.
vancouver scale scars (basal) | 0 day
  designed to evaluate the functional and aesthetic aspect of the scar. It consists of items related to pigmentation, vascularity, flexibility and height of the scar; the final score ranges from 0 to 13, with the lowest score corresponding to the best result. In the project in question will be used in the evaluation of the scar the items: vascularization, flexibility and height of the scar. It will be applied by a trained professional familiar with the use of the scale, according to the intervals established for the other evaluation instruments (zero and sequential evaluation after 45 and 90 days). This professional will evaluate and record the values corresponding to each of the scores mentioned below and in the end sum all the values generating a final score. The data will go to an envelope that will be sealed and opened at the end of the data collection.
vancouver scale scars (45o. day) | 45 days
  designed to evaluate the functional and aesthetic aspect of the scar. It consists of items related to pigmentation, vascularity, flexibility and height of the scar; the final score ranges from 0 to 13, with the lowest score corresponding to the best result. In the project in question will be used in the evaluation of the scar the items: vascularization, flexibility and height of the scar. It will be applied by a trained professional familiar with the use of the scale, according to the intervals established for the other evaluation instruments (zero and sequential evaluation after 45 and 90 days). This professional will evaluate and record the values corresponding to each of the scores mentioned below and in the end sum all the values generating a final score. The data will go to an envelope that will be sealed and opened at the end of the data collection.
vancouver scale scars (90o. day) | 90 days
  designed to evaluate the functional and aesthetic aspect of the scar. It consists of items related to pigmentation, vascularity, flexibility and height of the scar; the final score ranges from 0 to 13, with the lowest score corresponding to the best result. In the project in question will be used in the evaluation of the scar the items: vascularization, flexibility and height of the scar. It will be applied by a trained professional familiar with the use of the scale, according to the intervals established for the other evaluation instruments (zero and sequential evaluation after 45 and 90 days). This professional will evaluate and record the values corresponding to each of the scores mentioned below and in the end sum all the values generating a final score. The data will go to an envelope that will be sealed and opened at the end of the data collection.

CONTACTS AND LOCATIONS:
Overall Officials: Ana B Albuquerqu, master, Study Chair — Fernando Fiqueira IMI; Cláudia F Lima, doctorate, Study Chair — Hospital da Restauração Governador Paulo Guerra - Hospital da Restauração; Juliana N Maia, doctorate, Study Chair — Universidade Federal de Pernambuco - UFPE; Edlene L Ribeiro, doctorate, Study Chair — Fundação Oswaldo Cruz - Instituto Aggeu Magalhães
Locations (1):
- Alex Sandro Roland de Souza, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No